CLINICAL TRIAL: NCT02014584
Title: A Prospective Study of Sexual Function in Men Taking Dutasteride for the Treatment of Androgenetic Alopecia
Brief Title: Sexual Function in Men Receiving Dutasteride for Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200209
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Alopecia
Keywords: quality of life; safety; sexual function; male pattern hair loss (MPHL); Androgenic alopecia (AGA); dutasteride; satisfaction with hair growth
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dutasteride Arm (Experimental): Subjects will receive dutasteride 0.5 milligrams (mg) administered orally once daily for 24 Weeks
  Interventions: Drug: Dutasteride
- Placebo Arm (Placebo Comparator): Subjects will receive placebo administered orally once daily for 24 Weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — Dutasteride will be supplied as soft gelatin capsules, containing 0.5 mg of dutasteride to be administered orally.
  Arms: Dutasteride Arm
Drug: Placebo — Dutasteride matching placebo will be supplied as capsules to be administered orally.
  Arms: Placebo Arm

SUMMARY:
Treatment of male pattern hair loss (MPHL) or androgenetic alopecia (AGA) with 5α-reductase inhibitor (5-ARIs) has been associated with sexual dysfunction including erectile dysfunction and loss of libido. This will be a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the impact of dutasteride treatment on sexual function as well as subject satisfaction with hair growth and quality of life in men with AGA. This study will consist of a Screening Visit, a 4-week Placebo Run-in Phase, a Treatment Phase of 48 weeks, and a subsequent Follow-up Visit after 4 weeks. The treatment phase will include 24 weeks of double-blind, placebo controlled treatment and 24 weeks of open-label treatment with dutasteride. An extended 6-month Follow-up Visit will be conducted for any individuals with a change in erectile function at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject agrees to participate in the study and has signed and dated the informed consent form prior to the initiation of any study-related activities.
* AGA classified utilizing the Norwood-Hamilton classification.
* Men 18 to 50 years old, inclusively.
* Fluent and literate in local language with the ability to comprehend and record information on the International Index of Erectile Function, Hair Growth Satisfaction Scale, and DLQI questionnaires.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase and bilirubin ≤1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Have been in a stable heterosexual relationship during the last 6 months prior to screening and expect to maintain that relationship throughout the study.
* Must be sexually active: a man is considered sexually active if he has engaged in sexual intercourse (at least once) during the 4 weeks prior to screening.
* Men with a female partner of childbearing potential must agree to avoid exposure of his partner to semen by using a condom. Use of a condom must be from 2 weeks prior to administration of the first dose of study treatment until at least 5 half-lives for the drug (45 days) plus 3 months (i.e., a total of 4.5 months) to allow clearance of any residual drug in the semen after the last dose of study treatment.
* Willing to comply with study requirements.

Exclusion Criteria:

* Current or pre-existing sexual dysfunction as determined by: History of erectile dysfunction defined as the consistent inability to achieve or maintain an erection sufficient to permit satisfactory sexual intercourse. Score of ≤25 on the erectile function domain (IIEF-EF) of the IIEF at screening or at the baseline visit.
* Evidence of hypogonadism.
* Have a communicable skin or sexually-transmitted disease, or any rash or lesions on the penis or in the surrounding area (as reported by subject and evaluated by investigator).
* Serum prostate-specific antigen (PSA) >2.0 ng/mL at screening.
* Serum creatinine >1.5xULN at screening.
* Unstable liver disease (chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria).
* History of malignancy (including prostate cancer) within the past 5 years, except basal cell or squamous cell carcinoma of the skin.
* History of prostate cancer before the age of 50 years in a first degree relative.
* History of breast cancer or clinical breast examination suggestive of malignancy.
* Any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to screening; and uncontrolled diabetes or peptic ulcer disease that is uncontrolled by medical management.
* History or current evidence of any serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions that could, in the opinion of the investigator or the medical monitor, interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.Note: the investigator may consult with the GSK medical monitor if a condition could interfere with the subject's safety.
* Global scalp hair thinning, including occipital areas.
* Scarring of the scalp, including prior hair transplant or scalp reduction, or any other condition or disease of the scalp or hair, including diseases of the hair shaft (e.g., tinea infection, non-androgenetic-cause of alopecia, psoriatic dermatitis or other psoriatic lesions, or uncontrolled seborrheic dermatitis).
* History of hair transplantation at any time to correct AGA or use of hair weaving within 6 months prior to screening.
* History or evidence of hair loss other than AGA (e.g., due to an auto-immune, endocrine, mechanical or infectious process, or secondary to a scalp dermatological disorder).
* Use of any cosmetic product aimed at improving or correcting the signs of hair loss (e.g., scalp preparations with claims aiming at improved hair growth) within 2 weeks prior to screening.
* Use of light or laser treatments on the scalp (e.g., light emitting diode [LED] lamps) within 3 months prior to screening.
* Hypersensitivity to any 5-alpha reductase inhibitor (5-ARI) or its components or excipients or drugs chemically related to the study treatment.
* Use of dutasteride within 10 months prior to screening or use of finasteride within 6 months prior to screening.
* Previous use of systemic cytotoxic agents.
* Use of glucocorticoids (inhaled glucocorticoids are allowed; topical corticosteroids are allowed provided that they are not used on the scalp) within 3 months prior to screening.
* Use of the following prior to Baseline (within 1 week for topical products; within

  1 week or 5 half-lives, whichever is longer, for systemic treatments): Phosphodiesterase type 5 (PDE5) inhibitors (e.g., sildenafil, tadalafil, vardenafil); Minoxidil (oral or topical); Carpronium chloride; Systemic drugs with anti-androgenic properties (e.g., cyproterone acetate, spironolactone, ketoconazole, flutamide, and bicalutamide); Topical or systemic estrogen or progesterone; Drugs potentially causing hypertrichosis (e.g., cyclosporine, diazoxide, phenytoin, psoralens); Drugs potentially causing hypertrichosis or telogen effluvium (e.g., valproic acid); Anabolic steroids;
* Participation in any study of an investigational or marketed drug (within 5 half lives of drug) or device that may affect hair growth or sexual function prior to screening for this study. Note: Subject must not participate in any other drug or device studies during the course of this study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2016-03-19 (Actual); Study Completion 2016-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- GSK Investigational Site, Singapore, Singapore
- South Korea (9):
  - GSK Investigational Site, Chungcheongnam-do
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju-si, Jeollabuk-do
  - GSK Investigational Site, Kangwon-Do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a Screening Visit, a 4-week Placebo Run-in Period, a 24-week Double-Blind (DB) Treatment Period, followed by a 24-week Open-Label (OL) Active Treatment Period, and a 4-week post-treatment Follow-Up Visit.
Pre-assignment Details: Participants with an ongoing AE related to sexual function at the end of the treatment Period and participants who discontinued study treatment due to an AE related to sexual function entered a Targeted Follow-Up Period lasting until 24 weeks after the last dose of study treatment or until resolution of the sexual AE, whichever occurred first.
Groups:
- Placebo: Participants received placebo administered orally once daily for 24 weeks.
- Dutasteride 0.5 mg: Participants received dutasteride 0.5 mg administered orally once daily for 24 weeks.
- Placebo (DB)/Dutasteride 0.5 mg (OL): During double-blind treatment period participants received placebo administered orally once daily for 24 weeks. All participants completing the first 24-week treatment period received dutasteride 0.5 mg once daily for the second 24-week treatment period.
- Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL): During double-blind treatment period, participants received dutasteride 0.5 mg administered orally once daily for 24 weeks. All participants completing the first 24-week treatment period continued to receive dutasteride 0.5 mg once daily for the second 24-week treatment period.
- Targeted F/U: Placebo (DB)/Dutasteride 0.5 mg (OL): Participants with an ongoing AE related to sexual function at the end of the treatment Period and participants who discontinued study treatment due to an AE related to sexual function entered a Targeted Follow-Up Period (no study treatment administered) lasting until 24 weeks after the last dose of study treatment or until resolution of the sexual AE, whichever occurred first.
- Targeted F/U: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL): Participants with an ongoing AE related to sexual function at the end of the treatment Period and participants who discontinued study treatment due to an AE related to sexual function entered a Targeted Follow-Up Period (no study drug administered) lasting until 24 weeks after the last dose of study treatment or until resolution of the sexual AE, whichever occurred first.
Period: Double-Blind Period (24 Weeks)
Arm/Group | Placebo | Dutasteride 0.5 mg | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) | Targeted F/U: Placebo (DB)/Dutasteride 0.5 mg (OL) | Targeted F/U: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Started | 59 | 58 | 0 | 0 | 0 | 0
Completed | 57 | 52 | 0 | 0 | 0 | 0
Not Completed | 2 | 6 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0 | 0 | 0 | 0
Period: Open-Label Period (24 Weeks)
Arm/Group | Placebo | Dutasteride 0.5 mg | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) | Targeted F/U: Placebo (DB)/Dutasteride 0.5 mg (OL) | Targeted F/U: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Started | 0 | 0 | 49 | 48 | 0 | 0
Completed | 0 | 0 | 44 | 47 | 0 | 0
Not Completed | 0 | 0 | 5 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 0 | 0
Period: Target Follow-up (F/U) Period (24 Weeks)
Arm/Group | Placebo | Dutasteride 0.5 mg | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) | Targeted F/U: Placebo (DB)/Dutasteride 0.5 mg (OL) | Targeted F/U: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Started | 0 | 0 | 0 | 0 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dutasteride 0.5 mg | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (6.77) | 39.1 (6.65) | 39.0 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 59 | 58 | 117
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 49 | 48 | 97
  Asian - Southeast Asian Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) Related to Sexual Function in the Double-blind Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs related to sexual function are defined as: altered (decreased) libido, impotence, and ejaculation disorders.
Time Frame: 24 weeks
Population: Safety Population: all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants | 5 | 9
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.27, Fisher's Exact Test; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [-4.7 to 18.8]

2. Primary Outcome: Number of Participants With AE Related to Sexual Function in the Open-label Treatment Period
Description: as for outcome 1
Time Frame: 24 weeks
Population: Open-Label Period Population: all participants who entered the open-label period.
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants | 3 | 2

3. Primary Outcome: Number of Participants With AE Related to Sexual Function for the Double-blind and Open-label Combined Periods
Description: as for outcome 1
Time Frame: 48 weeks
Population: Dutasteride DB/OL Combined: all participants who entered the OL Period and taken Dutasteride in both the DB and the OL periods.
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 48
Participants | 10

4. Secondary Outcome: Duration and Persistence of AEs Related to Sexual Function in the Double-blind Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs related to sexual function are defined as: altered (decreased) libido, impotence, and ejaculation disorders. Duration is the total number of non-overlapping days for all events per subject. A duration is censored if there is at least one event with unknown start date or end date, in which case the censored duration is the minimum number of days that a subject has experienced any of these events. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). NA=not applicable.
Time Frame: 24 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Days
  Altered (decreased) libido n=2,1 | 88.5 (103.94) | 44.0 (NA) — The standard deviation was not calculated as only 1 participant was analyzed.
  Impotence, n=3, 7 | 68.3 (73.35) | 78.6 (83.09)
  Ejaculation disorder, n=0, 1 | NA (NA) — The mean and standard deviation was not calculated as no participants were analyzed. | 63.0 (NA) — The standard deviation was not calculated as only 1 participant was analyzed.

5. Secondary Outcome: Duration and Persistence of AEs Related to Sexual Function in the Open-label Treatment Period
Description: as for outcome 4
Time Frame: 24 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Days
  Altered (decreased) libido n=2,1 | 77.5 (71.42) | 135.0 (NA) — The standard deviation was not calculated as only 1 participant was analyzed.
  Impotence, n=1, 1 | 181.0 (NA) — The mean and standard deviation was not calculated as only 1 participant was analyzed. | 176.0 (NA) — The standard deviation was not calculated as only 1 participant was analyzed.
  Ejaculation disorder, n=0, 0 | NA (NA) — The mean and standard deviation was not calculated as no participants were analyzed. | NA (NA) — The mean and standard deviation was not calculated as no participants were analyzed.

6. Secondary Outcome: Duration and Persistence of AEs Related to Sexual Function in the Double-blind and Open-label Combined Periods
Description: as for outcome 4
Time Frame: 48 weeks
Population: Dutasteride DB/OL Combined population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 48
Days
  Altered (decreased) libido n=1 | 135.0 (NA) — The standard deviation was not calculated as only 1 participant was analyzed.
  Impotence, n=8 | 90.8 (84.28)
  Ejaculation disorder, n=1 | 63.0 (NA) — The standard deviation was not calculated as only 1 participant was analyzed.

7. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AEs Related to Sexual Function in the Double-blind Treatment Period
Description: as for outcome 1
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants | 0 | 0

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AEs Related to Sexual Function in the Open-label Treatment Period
Description: as for outcome 1
Time Frame: 24 weeks
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AEs Related to Sexual Function in the Double-blind and Open-label Combined Periods
Description: as for outcome 1
Time Frame: 48 weeks
Population: Dutasteride DB/OL Combined population
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 48
Participants | 0

10. Secondary Outcome: Number of Participants With AEs, Serious AEs (SAEs) and Possible Suicidality Related Adverse Events (PSRAEs) in the Double-blind Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment, all events of possible drug-induced liver injury with hyperbilirubinemia, breast cancer in male participants, or spontaneous abortion in female partner of male participant. The PSRAE form was used in this study to collect detailed information on the circumstances of reported AEs which, in the investigator's opinion, were possibly suicidality-related.
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  Any AE | 18 | 19
  Any SAE | 1 | 1
  PSRAE | 0 | 0

11. Secondary Outcome: Number of Participants With AEs, SAEs and PSRAEs in the Open-label Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.. SAE is defined as any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment, all events of possible drug-induced liver injury with hyperbilirubinemia, breast cancer in male participants, or spontaneous abortion in female partner of male participant. The PSRAE form was used in this study to collect detailed information on the circumstances of reported AEs which, in the investigator's opinion, were possibly suicidality-related.
Time Frame: 24 weeks
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  Any AE | 13 | 15
  Any SAE | 1 | 0
  PSRAE | 0 | 0

12. Secondary Outcome: Number of Participants With AEs, SAEs and PSRAEs in the Double-blind and Open-label Combined Periods
Description: as for outcome 11
Time Frame: 48 weeks
Population: Dutasteride DB/OL Combined population
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 48
Participants
  Any AE | 25
  Any SAE | 1
  PSRAE | 0

13. Secondary Outcome: Number of Participants With Treatment-related AEs in the Double-blind Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment related AE included events which the investigator classified as having a reasonable possibilty of being caused by the investigational product or whose classification was missing.
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants | 5 | 11

14. Secondary Outcome: Number of Participants With Treatment-related AEs in the Open-label Treatment Period
Description: as for outcome 13
Time Frame: 24 weeks
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants | 4 | 2

15. Secondary Outcome: Number of Participants With Treatment-related AEs in the Double-blind and Open-label Combined Periods
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment related AE included events which the investigator classified as having a reasonable possibility of being caused by the investigational product or whose classification was missing.
Time Frame: 48 weeks
Population: Dutasteride DB/OL Combined population
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 48
Participants | 11

16. Secondary Outcome: Number of Participants With AEs of Special Interest in the Double-blind Treatment Period
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs of special interest included those of sexual function: breast disorders (breast enlargement and breast tenderness), prostate cancer, cardiovascular events, and possible suicidality-related AEs (PSRAEs). Infrequent AEs of special interest included breast cancer, allergic reactions, depressed mood, hair changes, interference with formation of external genitalia in a male fetus, potential for decreased male fertility, and testicular pain and swelling. Special interest AEs are groups of MedDRA terms which have been defined in the analysis plan.
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  Altered (decreased libido) | 2 | 1
  Impotence | 3 | 7
  Ejaculation disorders | 0 | 1
  Breast disorder | 0 | 0
  Prostate cancer | 0 | 0
  Cardiovascular adverse event | 0 | 0
  Infrequent adverse events | 0 | 1

17. Secondary Outcome: Number of Participants With AEs of Special Interest in the Open-label Treatment Period
Description: as for outcome 16
Time Frame: 24 weeks
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  Altered (decreased libido) | 2 | 1
  Impotence | 1 | 1
  Ejaculation disorders | 0 | 0
  Breast disorder | 0 | 0
  Prostate cancer | 0 | 0
  Cardiovascular adverse event | 0 | 0
  Infrequent adverse events | 0 | 1

18. Secondary Outcome: Number of Participants With AEs of Special Interest in the Double-blind and Open-label Combined Periods
Description: as for outcome 16
Time Frame: 48 weeks
Population: Dutasteride DB/OL Combined population
Measure: Number; unit: Participants
Arm/Group | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 48
Participants
  Altered (decreased libido) | 1
  Impotence | 8
  Ejaculation disorders | 1
  Breast disorder | 0
  Prostate cancer | 0
  Cardiovascular adverse event | 0
  Infrequent adverse events | 2

19. Secondary Outcome: Suicidality Assessment Score by Using the Columbia Suicide Severity Rating Scale (C-SSRS) in the Double-blind Treatment Period
Description: Assessment of suicidality were done through use of the Columbia Suicide Severity Rating Scale (C-SSRS) for suicidal ideation with the ratings 1 to 5 (1. wish to be dead, 2. Non-specific suicidal thoughts, 3..without intent, 4. with intent but no plan, 5. with plan and intent) and for suicidal behavior with the ratings 6 to 9 (6.Prep acts/behavior, 7.aborted attempt, 8. interrupted attempt and 9. actual attempt). C-SSRS was administered at Day 1, Week 12, Week 24, and the early withdrawal visit if applicable .
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  Wish to be dead | 0 | 0
  Non-specific suicidal thoughts | 0 | 0
  Without intent | 0 | 0
  With intent but no plan | 0 | 0
  With plan and intent | 0 | 0
  Prep acts/behavior | 0 | 0
  Aborted attempt | 0 | 0
  Interrupted attempt | 0 | 0
  Actual attempt | 0 | 0
  Non-suicidal self injury behavior | 0 | 0

20. Secondary Outcome: Suicidality Assessment Score by Using the Columbia Suicide Severity Rating Scale (C-SSRS) in the Open-label Treatment Period
Description: Assessment of suicidality were done through use of the Columbia Suicide Severity Rating Scale (C-SSRS) for suicidal ideation with the ratings 1 to 5 (1. wish to be dead, 2. Non-specific suicidal thoughts, 3. without intent, 4. with intent but no plan, 5. with plan and intent) and for suicidal behavior with the ratings 6 to 9 (6.Prep acts/behavior, 7.aborted attempt, 8. interrupted attempt and 9. actual attempt). C-SSRS was administered at Day 1, Week 12, Week 24, and the early withdrawal visit if applicable .
Time Frame: 24 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  Wish to be dead | 0 | 0
  Non-specific suicidal thoughts | 0 | 0
  Without intent | 0 | 0
  With intent but no plan | 0 | 0
  With plan and intent | 0 | 0
  Prep acts/behavior | 0 | 0
  Aborted attempt | 0 | 0
  Interrupted attempt | 0 | 0
  Actual attempt | 0 | 0
  Non-suicidal self injury behavior | 0 | 0

21. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in the Double-blind Treatment Period
Description: The Baseline blood presssure assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 12 and Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
millimeter of mercury (mmHg)
  SBP Week 12, n=59, 53 | 0.9 (9.71) | -0.1 (10.46)
  SBP Week 24, n=57, 52 | -1.0 (13.27) | -2.0 (14.08)
  DBP Week 12, n=59, 53 | 2.1 (7.99) | 1.6 (9.23)
  DBP Week 24, n=57, 52 | -0.2 (9.78) | -1.5 (9.73)

22. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure in the Open-label Treatment Period
Description: Baseline blood presure assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 12 and Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
mmHg
  SBP Week 12, n=46, 48 | -0.9 (10.02) | 0.1 (12.76)
  SBP Week 24, n=44, 47 | -0.7 (11.30) | 0.4 (12.90)
  DBP Week 12, n=46, 48 | -0.8 (8.87) | -0.6 (9.00)
  DBP Week 24, n=44, 47 | -1.4 (8.26) | 0.9 (11.23)

23. Secondary Outcome: Change From Baseline in Heart Rate in the Double-blind Treatment Period
Description: The Baseline heart rate assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 12 and Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Beats per Minute
  Week 12, n=59, 53 | 0.3 (8.19) | -0.6 (11.39)
  Week 24, n=57, 52 | 0.6 (9.21) | -0.7 (11.20)

24. Secondary Outcome: Change From Baseline in Heart Rate in the Open-label Treatment Period
Description: Baseline heart rate assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 12 and Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Beats per Minute
  Week 12, n=46, 48 | -1.5 (10.86) | 1.1 (13.15)
  Week 24, n=44, 47 | -0.3 (10.83) | 1.2 (11.26)

25. Secondary Outcome: Number of Participants With Frequency of Systolic and Diastolic Blood Pressure of Clinical Concern in the Double-blind Treatment Period
Description: The Baseline blood presssure assessment was defined as the latest assessment on or before the double-blind treatment start. The clinical concern range for vital signs was defined as: Systolic blood pressure (lower: <80, upper: >165) and diastolic blood pressure: (lower: <40, upper: >105).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  Baseline SBP <80 mmHg | 0 | 0
  Baseline SBP >165 mmHg | 0 | 0
  Baseline DBP <40 mmHg | 0 | 0
  Baseline DBP >105 mmHg | 0 | 0
  Post Baseline SBP <80 mmHg | 0 | 0
  Post Baseline SBP >165 mmHg | 0 | 0
  Post Baseline DBP <40 mmHg | 0 | 0
  Post Baseline DBP >105 mmHg | 1 | 2

26. Secondary Outcome: Number of Participants With Frequency of Systolic and Diastolic Blood Pressure of Clinical Concern in the Open-label Treatment Period
Description: The Baseline blood presssure assessment was defined as the latest assessment on or before the open-label treatment start. The clinical concern range for vital signs was defined as: systolic blood pressure (lower: <80, upper: >165) and diastolic blood pressure: (lower: <40, upper: >105).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  Baseline SBP <80 mmHg | 0 | 0
  Baseline SBP >165 mmHg | 0 | 0
  Baseline DBP <40 mmHg | 0 | 0
  Baseline DBP >105 mmHg | 0 | 0
  Post Baseline SBP <80 mmHg | 0 | 0
  Post Baseline SBP >165 mmHg | 0 | 0
  Post Baseline DBP <40 mmHg | 0 | 0
  Post Baseline DBP >105 mmHg | 0 | 0

27. Secondary Outcome: Number of Participants With Frequency of Heart Rate of Clinical Concern in the Double-blind Treatment Period
Description: The Baseline heart rate assessment was defined as the latest assessment on or before the double-blind treatment start. The clinical concern range for heart rate was defined as: (lower: <40, upper: >100).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  Baseline <40 | 0 | 0
  Baseline >100 | 1 | 1
  Post- Baseline <40 | 0 | 0
  Post- Baseline >100 | 1 | 2

28. Secondary Outcome: Number of Participants With Frequency of Heart Rate of Clinical Concern in the Open-label Treatment Period
Description: Baseline heart rate assessment was defined as the latest assessment on or before the open-label treatment start. The clinical concern range for heart rate was defined as: (lower: <40, upper: >100).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  Baseline <40 | 0 | 0
  Baseline >100 | 1 | 1
  Post- Baseline <40 | 0 | 0
  Post- Baseline >100 | 3 | 5

29. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameters in the Double-blind Treatment Period
Description: Hematology parameters included: platelet count, white blood cell (WBC) count, basophils, eosinophils, lymphocytes, monocytes, segmented neutrophils and total neutrophils at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga per Liter (GI/L)
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Giga per Liter (GI/L)
  Platelet Count DB Week 24, n=54, 47 | 2.2 (37.79) | 9.6 (24.01)
  Platelet Count Final Value, n=55, 48 | 2.3 (37.45) | 9.0 (23.93)
  WBC DB Week 24, n=55, 51 | 0.1 (1.39) | 0.1 (1.32)
  WBC Final Value, n=56, 52 | 0.1 (1.35) | 0.1 (1.16)
  Basophils DB Week 24, n=50, 46 | -0.0 (0.03) | -0.0 (0.03)
  Basophils Final Value, n=51, 47 | -0.0 (0.03) | -0.0 (0.03)
  Eosinophils DB Week 24, n=50, 46 | -0.0 (0.15) | -0.0 (0.11)
  Eosinophils Final Value, n=51, 47 | -0.0 (0.15) | -0.0 (0.13)
  Lymphocytes DB Week 24, n=50, 46 | 0.0 (0.76) | -0.1 (0.59)
  Lymphocytes Final Value, n=51, 47 | 0.1 (0.75) | -0.0 (0.59)
  Monocytes DB Week 24, n=50, 46 | 0.0 (0.16) | -0.0 (0.13)
  Monocytes Final Value, n=51, 47 | 0.0 (0.16) | -0.0 (0.13)
  Segmented Neutrophils DB Week 24, n=50, 46 | 0.1 (1.27) | 0.2 (1.31)
  Segmented Neutrophils Final Value, n=51, 47 | 0.1 (1.26) | 0.2 (1.14)
  Total Neutrophils DB Week 24, n=50, 46 | 0.1 (1.27) | 0.2 (1.31)
  Total Neutrophils Final Value, n=51, 47 | 0.1 (1.26) | 0.2 (1.14)

30. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameters in the Open-label Treatment Period
Description: Hematology parameters included: platelet count, white blood cell (WBC) count, basophils, eosinophils, lymphocytes, monocytes, segmented neutrophils, and total neutrophils at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: Giga per Liter (GI/L)
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Giga per Liter (GI/L)
  Platelet Count OL Week 24, n=42, 45 | 2.1 (30.41) | -2.5 (19.83)
  Platelet Count Final Value, n=42, 45 | 2.1 (30.41) | -3.4 (20.33)
  WBC OL Week 24, n=42, 47 | 0.2 (1.23) | 0.2 (1.71)
  WBC Final Value, n=42, 47 | 0.1 (1.25) | 0.1 (1.68)
  Basophils OL Week 24, n=39, 44 | -0.0 (0.02) | 0.0 (0.02)
  Basophils Final Value, n=40, 44 | -0.0 (0.02) | 0.0 (0.02)
  Eosinophils OL Week 24, n=39, 44 | -0.0 (0.17) | 0.0 (0.14)
  Eosinophils Final Value, n=40, 44 | -0.0 (0.17) | 0.0 (0.14)
  Lymphocytes OL Week 24, n=39, 44 | -0.0 (0.47) | 0.1 (0.50)
  Lymphocytes Final Value, n=40, 44 | -0.0 (0.46) | 0.1 (0.50)
  Monocytes OL Week 24, n=39, 44 | -0.0 (0.12) | -0.0 (0.12)
  Monocytes Final Value, n=40, 44 | -0.0 (0.13) | -0.0 (0.12)
  Segmented Neutrophils OL Week 24, n=39, 44 | 0.2 (1.19) | 0.0 (1.72)
  Segmented Neutrophils Final Value, n=40, 44 | 0.2 (1.20) | 0.0 (1.72)
  Total Neutrophils OL Week 24, n=39, 44 | 0.2 (1.19) | 0.0 (1.72)
  Total Neutrophils Final Value, n=40, 44 | 0.2 (1.20) | 0.0 (1.72)

31. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameter in the Double-blind Treatment Period: Hematocrit
Description: Hematology parameter included: hematocrit at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of RBCs
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Proportion of RBCs
  DB Week 24, n=55, 51 | -0.0 (0.02) | 0.0 (0.02)
  Final Value, n=56, 52 | -0.0 (0.02) | 0.0 (0.02)

32. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameter in the Open-label Treatment Period: Hematocrit
Description: Hematology parameter included: hematocrit at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: Proportion of RBCs
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Proportion of RBCs
  OL Week 24, n=43, 47 | 0.0 (0.02) | 0.0 (0.02)
  Final Value, n=43, 47 | 0.0 (0.02) | 0.0 (0.02)

33. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameter in the Double-blind Treatment Period: Hemoglobin
Description: Hematology parameter included: hemoglobin at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
G/L
  DB Week 24, n=55, 51 | -2.0 (6.56) | -0.8 (5.33)
  Final Value, n=56, 52 | -2.0 (6.46) | -0.8 (5.68)

34. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameter in the Open-label Treatment Period: Hemoglobin
Description: Hematology parameters included: hemoglobin at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
G/L
  OL Week 24, n=43, 47 | -1.5 (7.65) | -1.4 (5.30)
  Final Value, n=43, 47 | -1.5 (7.65) | -1.4 (5.30)

35. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameter in the Double-blind Treatment Period: Red Blood Cell (RBC) Count
Description: Hematology parameter included: RBC at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: T/L
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
T/L
  DB Week 24, n=55, 51 | -0.0 (0.25) | 0.0 (0.20)
  Final Value, n=56, 52 | -0.0 (0.25) | 0.0 (0.21)

36. Secondary Outcome: Change From Baseline in the Indicated Hematology Parameter in the Open-label Treatment Period: Red Blood Cell (RBC) Count
Description: Hematology parameter included: RBC at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: T/L
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
T/L
  OL Week 24, n=43, 47 | -0.1 (0.27) | -0.1 (0.20)
  Final Value, n=43, 47 | -0.1 (0.27) | -0.1 (0.20)

37. Secondary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters in the Double-blind Treatment Period: Albumin and Total Protein
Description: Clinical chemistry parameters included: albumin and total protein at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
G/L
  Albumin, DB Week 24, n=57, 52 | 0.2 (1.82) | -0.1 (2.15)
  Albumin, Final Value, n=58, 53 | 0.2 (1.81) | -0.1 (2.21)
  Total Protein, DB Week 24, n=57, 52 | -0.1 (3.14) | -0.0 (3.64)
  Total Protein, Final Value, n=58, 53 | -0.1 (3.09) | 0.1 (3.79)

38. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters in the Open-label Treatment Period: Albumin and Total Protein
Description: as for outcome 37
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
G/L
  Albumin OL Week 24, n=44, 47 | -0.6 (2.02) | -1.1 (2.02)
  Albumin Final Value, n=44, 47 | -0.5 (2.05) | -1.1 (2.02)
  Total Protein OL Week 24, n=44, 47 | -0.8 (3.90) | -2.4 (3.23)
  Total Protein Final Value, n=44, 47 | -0.7 (3.94) | -2.4 (3.23)

39. Secondary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters in the Double-blind Treatment Period
Description: Clinical chemistry parameters included: alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST) and gamma glutamyl transferase (GGT) at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
IU/L
  ALT DB Week 24, n=57, 52 | 0.9 (21.69) | 4.0 (12.70)
  ALT Final Value, n=58, 53 | 1.0 (21.51) | 3.5 (12.37)
  ALP DB Week 24, n=57, 52 | -4.8 (10.41) | -4.1 (8.16)
  ALP Final Value, n=58, 53 | -4.8 (10.35) | -4.5 (8.82)
  AST DB Week 24, n=57, 51 | 0.7 (10.42) | 0.5 (6.99)
  AST Final Value, n=58, 52 | 0.6 (10.34) | 0.3 (6.65)
  GGT DB Week 24, n=57, 52 | -6.4 (30.95) | -1.1 (15.84)
  GGT Final Value, n=58, 53 | -6.3 (30.69) | -1.1 (15.67)

40. Secondary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters in the Open-label Treatment Period
Description: Clinical chemistry parameters included: ALT, ALP, AST, and GGT at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
IU/L
  ALT OL Week 24, n=44, 47 | -1.4 (19.22) | -1.7 (13.07)
  ALT Final Value, n=44, 47 | -1.3 (19.25) | -1.7 (13.07)
  ALP OL Week 24, n=44, 47 | 0.0 (9.87) | -3.3 (7.59)
  ALP Final Value, n=44, 47 | 0.0 (9.85) | -3.3 (7.59)
  AST OL Week 24, n=43, 47 | -0.2 (7.00) | 0.1 (8.90)
  AST Final Value, n=44, 47 | -0.5 (7.18) | 0.1 (8.90)
  GGT OL Week 24, n=44, 47 | 3.7 (13.13) | 0.6 (19.59)
  GGT Final Value, n=44, 47 | 3.7 (13.13) | 0.6 (19.59)

41. Secondary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters in the Double-blind Treatment Period: Creatinine, Direct Bilirubin and Total Bilirubin
Description: Clinical chemistry parameters included: creatinine, direct bilirubin, total bilirubin at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: UMOL/L
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
UMOL/L
  Creatinine DB Week 24, n=57, 52 | 1.7 (8.20) | -0.7 (9.41)
  Creatinine Final Value, n=58, 53 | 1.6 (8.12) | -0.8 (9.37)
  Direct bilirubin DB Week 24, n=57, 52 | -0.2 (0.86) | -0.3 (0.93)
  Direct bilirubin Final Value, n=58, 53 | -0.1 (0.90) | -0.2 (0.93)
  Total bilirubin DB Week 24, n=57, 52 | -1.1 (4.66) | -1.1 (4.56)
  Total bilirubin Final Value, n=58, 53 | -1.1 (4.65) | -1.0 (4.36)

42. Secondary Outcome: Change From Baseline in the Clinical Chemistry Parameters in the Open-label Treatment Period: Creatinine, Direct Bilirubin and Total Bilirubin.
Description: Clinical chemistry parameters included: creatinine, direct bilirubin, total bilirubin at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: UMOL/L
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
UMOL/L
  Creatinine OL Week 24, n=44, 47 | 1.1 (12.01) | -0.2 (6.66)
  Creatinine Final Value, n=44, 47 | 1.2 (12.01) | -0.2 (6.66)
  Direct bilirubin OL Week 24, n=44, 47 | 0.1 (0.89) | 0.1 (1.02)
  Direct bilirubin Final Value, n=44, 47 | 0.1 (0.90) | 0.1 (1.02)
  Total bilirubin OL Week 24, n=44, 47 | 0.9 (3.84) | 0.4 (5.10)
  Total bilirubin Final Value, n=44, 47 | 1.0 (3.91) | 0.4 (5.10)

43. Secondary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters in the Double-blind Treatment Period: Glucose, Potassium, Sodium and Urea/Blood Urea Nitrogen (BUN)
Description: Clinical chemistry parameters included: glucose, potassium, sodium, and urea/BUN at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the double-blind treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: MMOL/L
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
MMOL/L
  Glucose DB Week 24, n=57, 52 | 0.1 (1.58) | 0.0 (0.36)
  Glucose Final Value, n=58, 53 | 0.1 (1.57) | 0.0 (1.18)
  Potassium DB Week 24, n=57, 51 | 0.0 (0.32) | 0.0 (0.29)
  Potassium Final Value n=58, 52 | 0.0 (0.32) | 0.0 (0.30)
  Sodium DB Week 24, n=57, 52 | 0.5 (1.60) | 0.2 (2.13)
  Sodium Final Value, n=58, 53 | 0.5 (1.61) | 0.4 (1.87)
  Urea/BUN Final Value, n=57, 52 | 0.2 (1.22) | 0.0 (1.32)
  Urea/BUN Value, n=58, 53 | 0.2 (1.23) | 0.1 (1.33)

44. Secondary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters in the Open-label Treatment Period: Glucose, Potassium, Sodium and Urea/BUN.
Description: Clinical chemistry parameters included: glucose, potassium, sodium, and urea/BUN at the indicated time points (Week 24 and final value). The Baseline assessment was defined as the latest assessment on or before the open-label treatment start. Change from Baseline is post-Baseline value minus Baseline value. A final value for each period is defined as the latest post-Baseline value available in the period. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: MMOL/L
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
MMOL/L
  Glucose OL Week 24, n=44, 47 | 0.3 (1.48) | 0.2 (1.13)
  Glucose Final Value, n=44, 47 | 0.3 (1.48) | 0.2 (1.13)
  Potassium OL Week 24, n=43, 47 | -0.1 (0.36) | -0.0 (0.30)
  Potassium Final Value, n=44, 47 | -0.0 (0.37) | -0.0 (0.30)
  Sodium OL Week 24, n=44, 47 | -0.9 (2.51) | -0.6 (1.79)
  Sodium Final Value, n=44, 47 | -0.9 (2.51) | -0.6 (1.79)
  Urea/BUN OL Week 24, n=44, 47 | 0.3 (1.50) | -0.1 (1.15)
  Urea/BUN Final Value, n=44, 47 | 0.3 (1.50) | -0.1 (1.15)

45. Secondary Outcome: Incidence of Premature Discontinuations in the Double-blind Treatment Period
Description: Participants were referred as premature discontinuations if they do not complete the double-blind period. The reasons for premature withdrawal were protocol deviation, lost to follow-up and withdrawal of consent by participants.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants | 2 | 6

46. Secondary Outcome: Incidence of Premature Discontinuations in the Open-label Treatment Period
Description: Participants were referred as premature discontinuations if they do not complete the open-label treatment period. The reasons for premature withdrawal were protocol deviation, lost to follow-up and withdrawal of consent by participants.
Time Frame: Week 48
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants | 5 | 1

47. Secondary Outcome: Number of Participants With a Change in Sexual Function Defined as a Negative Change From Baseline in the International Index of Erectile Function (IIEF) Erectile Function Domain (IIEF-EF) Score of >=4 Units in the Double-blind Treatment Period
Description: The IIEF is a validated 15-item questionnaire with individual items of the questionnaire assigned to five separate domains of sexual function (i.e., erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction). The IIEF was employed to assess treatment-related changes in men with erectile dysfunction. The erectile function domain of the IIEF (IIEF-EF) includes Questions 1 through 5 and Question 15 (maximum score of 30). A clinically meaningful gradient of severity of erectile dysfunction (ED) has been developed, indicating that a score of greater than 25 represents an individual without ED while men scoring <=25 may be classified as having ED. The values are presented for Week 4, Week 12 and Week 24. The Baseline assessment was defined as the latest assessment on or before the DB treatment start. Change from Baseline is post-Baseline value minus Baseline value.
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  DB Week 4 | 3 | 1
  DB Week 12 | 4 | 7
  DB Week 24 | 3 | 6
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.62, Fisher's Exact Test; Median Difference (Final Values) = -3.5, 95% CI 2-sided [-10.4 to 3.4] — DB Week 4
Statistical Analysis 2: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.34, Fisher's Exact Test; Median Difference (Final Values) = 6.4, 95% CI 2-sided [-4.7 to 17.6] — DB Week 12
Statistical Analysis 3: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.31, Fisher's Exact Test; Median Difference (Final Values) = 6.3, 95% CI 2-sided [-4.2 to 16.7] — DB Week 24

48. Secondary Outcome: Number of Participants With a Change in Sexual Function Defined as a Negative Change From Baseline in the IIEF Erectile Function Domain (IIEF-EF) Score of >=4 Units in the Open-label Treatment Period
Description: as for outcome 47
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: Open-Label Period Population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  OL Week 4 | 2 | 2
  OL Week 12 | 2 | 3
  OL Week 24 | 1 | 5

49. Secondary Outcome: Change From Baseline in Total Score of the IIEF in the Double-blind Treatment Period
Description: The IIEF is a validated 15-item questionnaire with individual items of the questionnaire assigned to five separate domains of sexual function (i.e., erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction). The IIEF was employed to assess treatment-related changes in men with erectile dysfunction. Overall score range is 0-75. The erectile function score range is 0-30, intercourse satisfaction score range is 0-15, orgasmic function score range is 0-10, sexual desire score range is 0-10, overall satisfaction score range is 0-10. A decrease from Baseline indicates a worsening. The change from Baseline values are presented for Week 4, Week 12 and Week 24. The Baseline assessment was defined as the latest assessment on or before the DB treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Scores on a Scale
  DB Week 4, n=56, 54 | -1.4 (0.56) | -0.0 (0.57)
  DB Week 12, n= 59, 53 | -0.9 (0.75) | -2.2 (0.79)
  DB Week 24, n=57, 51 | -1.2 (0.71) | -1.2 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.082, t-test from general linear model; Adjusted mean difference = 1.4, 95% CI 2-sided [-0.2 to 3.0], Standard Error of Mean 0.80 — DB Week 4
Statistical Analysis 2: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.25, t-test from general linear model; Adjusted mean difference = -1.3, 95% CI 2-sided [-3.4 to 0.9], Standard Error of Mean 1.09 — DB Week 12
Statistical Analysis 3: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.99, t-test from general linear model; Adjusted mean difference = 0.0, 95% CI 2-sided [-2.0 to 2.1], Standard Error of Mean 1.04 — DB Week 24

50. Secondary Outcome: Change From Baseline in Total Score of the IIEF in the Open-label Treatment Period
Description: as for outcome 49
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: Open-Label Period Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Scores on a Scale
  OL Week 4, n=47, 48 | 0.4 (5.55) | 0.2 (3.04)
  OL Week 12, n=46, 48 | -0.6 (5.28) | -0.3 (5.34)
  OL Week 24, n=44, 47 | -0.1 (5.73) | -2.6 (11.05)

51. Secondary Outcome: Change From Baseline in the Individual Domain Scores (Erectile Function, Orgasmic Function, Sexual Desire, Intercourse Satisfaction and Overall Sexual Satisfaction) of the IIEF in the Double-blind Treatment Period
Description: The IIEF is a validated 15-item questionnaire with individual items of the questionnaire assigned to five separate domains of sexual function (i.e., erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction). The IIEF was employed to assess treatment-related changes in men with erectile dysfunction. Overall score range is 0-75. The erectile function score range is 0-30, intercourse satisfaction score range is 0-15, orgasmic function score range is 0-10, sexual desire score range is 0-10, overall satisfaction score range is 0-10. A decrease from Baseline indicates a worsening. The Baseline assessment was defined as the latest assessment on or before the DB treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Scores on a Scale
  Erectile Function DB Week 4, n=56, 54 | -0.5 (0.23) | -0.3 (0.24)
  Erectile Function DB Week 12, n= 59, 53 | -0.5 (0.35) | -1.3 (0.37)
  Erectile Function DB Week 24, n=57, 52 | -0.5 (0.42) | -1.2 (0.44)
  Intercourse satisfaction DB Week 4, n=56, 54 | -0.3 (0.16) | 0.0 (0.16)
  Intercourse satisfaction DB Week 12, n=59, 53 | -0.1 (0.23) | -0.2 (0.24)
  Intercourse satisfaction DB Week 24, n=57, 52 | -0.3 (0.23) | -0.4 (0.24)
  Orgasmic function DB Week 4, n=56, 54 | -0.0 (0.11) | 0.1 (0.11)
  Orgasmic function DB Week 12, n=59, 53 | 0.0 (0.10) | -0.1 (0.11)
  Orgasmic function DB Week 24, n=57, 52 | -0.0 (0.15) | -0.1 (0.16)
  Sexual desire DB Week 4, n=56, 54 | -0.4 (0.14) | -0.1 (0.15)
  Sexual desire DB Week 12, n=59, 53 | -0.2 (0.15) | -0.4 (0.16)
  Sexual desire DB Week 24, n=57, 52 | -0.2 (0.18) | -0.2 (0.19)
  Overall sexual satisfaction DB Week 4, n=56, 54 | -0.1 (0.12) | 0.1 (0.12)
  Overall sexual satisfaction DB Week 12, n=59, 53 | -0.1 (0.13) | -0.2 (0.14)
  Overall sexual satisfaction DB Week 24, n=57, 51 | -0.1 (0.15) | -0.2 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.46, t-test from general linear model; Adjusted mean difference = 0.2, 95% CI 2-sided [-0.4 to 0.9], Standard Error of Mean 0.33 — Erectile Function DB Week 4
Statistical Analysis 2: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.14, t-test from general linear model; Adjusted mean difference = -0.8, 95% CI 2-sided [-1.8 to 0.3], Standard Error of Mean 0.52 — Erectile Function DB Week 12
Statistical Analysis 3: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.27, t-test from general linear model; Adjusted mean difference = -0.7, 95% CI 2-sided [-1.9 to 0.5], Standard Error of Mean 0.61 — Erectile Function DB Week 24
Statistical Analysis 4: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.13, t-test from general linear model; Adjusted mean difference = 0.3, 95% CI 2-sided [-0.1 to 0.8], Standard Error of Mean 0.23 — Intercourse satisfaction DB Week 4
Statistical Analysis 5: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.73, t-test from general linear model; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.33 — Intercourse satisfaction DB Week 12
Statistical Analysis 6: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.64, t-test from general linear model; Adjusted mean difference = -0.2, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.34 — Intercourse satisfaction DB Week 24
Statistical Analysis 7: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.23, t-test from general linear model; Adjusted mean difference = 0.2, 95% CI 2-sided [-0.1 to 0.5], Standard Error of Mean 0.16 — Orgasmic function DB Week 4
Statistical Analysis 8: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.33, t-test from general linear model; Adjusted mean difference = -0.2, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.15 — Orgasmic function DB Week 12
Statistical Analysis 9: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.64, t-test from general linear model; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.23 — Orgasmic function DB Week 24
Statistical Analysis 10: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.19, t-test from general linear model; Adjusted mean difference = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.21 — Sexual desire DB Week 4
Statistical Analysis 11: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.28, t-test from general linear model; Adjusted mean difference = -0.2, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.22 — Sexual desire DB Week 12
Statistical Analysis 12: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 1.00, t-test from general linear model; Adjusted mean difference = -0.0, 95% CI 2-sided [-0.5 to 0.5], Standard Error of Mean 0.27 — Sexual desire DB Week 24
Statistical Analysis 13: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.28, t-test from general linear model; Adjusted mean difference = 0.2, 95% CI 2-sided [-0.2 to 0.5], Standard Error of Mean 0.17 — Overall sexual satisfaction DB Week 4
Statistical Analysis 14: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.64, t-test from general linear model; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.20 — Overall sexual satisfaction DB Week 12
Statistical Analysis 15: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.69, t-test from general linear model; Adjusted mean difference = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.22 — Overall sexual satisfaction DB Week 24

52. Secondary Outcome: Change From Baseline in the Individual Domain Scores (Erectile Function, Orgasmic Function, Sexual Desire, Intercourse Satisfaction and Overall Sexual Satisfaction) of the IIEF in the Open-label Treatment Period
Description: The IIEF is a validated 15-item questionnaire with individual items of the questionnaire assigned to five separate domains of sexual function (i.e., erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction). The IIEF was employed to assess treatment-related changes in men with erectile dysfunction. Overall score range is 0-75. The erectile function score range is 0-30, intercourse satisfaction score range is 0-15, orgasmic function score range is 0-10, sexual desire score range is 0-10, overall satisfaction score range is 0-10. A decrease from Baseline indicates a worsening. The Baseline assessment was defined as the latest assessment on or before the OL treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: Open-label Period Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Scores on a Scale
  Erectile Function OL Week 4, n=47, 48 | 0.0 (2.30) | -0.1 (1.76)
  Erectile Function OL Week 12, n= 46, 48 | -0.1 (1.86) | -0.3 (2.99)
  Erectile Function OL Week 24, n=44, 47 | 0.0 (1.62) | -1.4 (5.22)
  Intercourse satisfaction OL Week 4, n=47, 48 | 0.1 (1.45) | 0.0 (1.03)
  Intercourse satisfaction OL Week 12, n= 46, 48 | -0.2 (1.57) | -0.1 (1.93)
  Intercourse satisfaction OL Week 24, n=44, 47 | -0.1 (1.93) | -0.5 (2.60)
  Orgasmic function OL Week 4, n=47, 48 | 0.1 (0.88) | 0.1 (0.65)
  Orgasmic function OL Week 12, n= 46, 48 | 0.0 (0.80) | -0.1 (0.56)
  Orgasmic function OL Week 24, n=44, 47 | 0.1 (0.80) | -0.4 (2.12)
  Sexual desire OL Week 4, n=47, 48 | 0.1 (1.50) | 0.0 (1.01)
  Sexual desire OL Week 12, n= 46, 48 | -0.2 (1.60) | -0.1 (1.07)
  Sexual desire OL Week 24, n=44, 47 | -0.0 (1.72) | -0.1 (1.04)
  Overall sexual satisfaction OL Week 4, n=47, 48 | 0.0 (1.13) | 0.1 (0.73)
  Overall sexual satisfaction OL Week 12, n= 46, 48 | -0.2 (0.99) | 0.2 (0.71)
  Overall sexual satisfaction OL Week 24, n=44, 47 | -0.2 (1.10) | -0.1 (1.45)

53. Secondary Outcome: Change From Baseline in Participant Satisfaction With Hair Growth as Assessed by the Total Score of the Hair Growth Satisfaction Scale (HGSS) in the Double-blind Treatment Period
Description: The HGSS assessed participants satisfaction with hair appearance and growth by scoring 5 questions on a 7-point scale ranging from 1=very dissatisfied to 7= very satisfied with a maximum score of 35. The Baseline assessment was defined as the latest assessment on or before the DB treatment start. Change from Baseline is post-Baseline value minus Baseline value. A decrease from Baseline indicates a worsening. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 12 and Week 24
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Scores on a Scale
  DB Week 12, n= 58, 53 | 1.3 (0.79) | 2.4 (0.82)
  DB Week 24, n=57, 52 | -0.1 (0.79) | 3.2 (0.82)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.33, t-test from general linear model; Adjusted mean difference = 1.1, 95% CI 2-sided [-1.1 to 3.4], Standard Error of Mean 1.14 — DB Week 12
Statistical Analysis 2: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.004, t-test from general linear model; Adjusted mean difference = 3.3, 95% CI 2-sided [1.1 to 5.6], Standard Error of Mean 1.14 — DB Week 24

54. Secondary Outcome: Change From Baseline in Participant Satisfaction With Hair Growth as Assessed by the Total Score of the HGSS in the Open-label Treatment Period
Description: The HGSS assessed participants satisfaction with hair appearance and growth by scoring 5 questions on a 7-point scale ranging from 1=very dissatisfied to 7=very satisfied with a maximum score of 35. The Baseline assessment was defined as the latest assessment on or before the OL treatment start. Change from Baseline is post-Baseline value minus Baseline value. A decrease from Baseline indicates a worsening. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline and up to Week 24
Population: Open-label Period Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 44 | 47
Scores on a Scale | 4.5 (6.96) | 4.5 (7.23)

55. Secondary Outcome: Change From Baseline in the Total Score of the Dermatology Life Quality Index (DLQI) in the Double-blind Treatment Period
Description: The DLQI was a 10-item questionnaire designed to evaluate the effect of skin conditions (alopecia) on the participants quality of life. Each item was scored on a 4-point scale ranging from 0 to 3 with a maximum score of 30. Higher scores represent greater impairment in quality of life. The Baseline assessment was defined as the latest assessment on or before the DB treatment start. Change from Baseline is post-Baseline value minus Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 12 and Week 24
Population: Safety Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Scores on a Scale
  DB Week 12, n= 58, 53 | 0.2 (0.35) | -0.4 (0.37)
  DB Week 24, n=57, 52 | 0.7 (0.52) | 0.2 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.22, t-test from general linear model; Adjusted mean difference = -0.6, 95% CI 2-sided [-1.7 to 0.4], Standard Error of Mean 0.51 — DB Week 12
Statistical Analysis 2: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.50, t-test from general linear model; Adjusted mean difference = -0.5, 95% CI 2-sided [-2.0 to 1.0], Standard Error of Mean 0.76 — DB Week 24

56. Secondary Outcome: Change From Baseline in the Total Score of the DLQI in the Open-label Treatment Period
Description: The DLQI was a 10-item questionnaire designed to evaluate the effect of skin conditions (alopecia) on the participants quality of life. Each item was scored on a 4-point scale ranging from 0 to 3 with a maximum score of 30. Higher scores represent greater impairment in quality of life. The Baseline assessment was defined as the latest assessment on or before the OL treatment start. Change from Baseline is post-Baseline value minus Baseline value.
Time Frame: Baseline and Upto Week 24
Population: Open-label Period Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Scores on a Scale | -1.0 (3.92) | -0.8 (3.77)

57. Secondary Outcome: Change From Baseline in Participants Perception of Sexual Function Measured by Responses to the Global Assessment Questions in the Double-blind Treatment Period
Description: The global assessment questions consist of 2 questions, recording how much the participant perceives his sexual life has changed and how he perceives his ability to achieve and maintain erections has changed, compared to how it was before he began receiving treatment in this study. The wording of these questions were based on the Patient Global Impression of Improvement questionnaire, which was validated for use in the assessment of improvement in stress urinary incontinence. The questions were scored on a 7-point scale.The Baseline assessment was defined as the latest assessment on or before the DB treatment start.
Time Frame: Baseline and up to Week 24
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 59 | 58
Participants
  Baseline, Erection ability, Very Much Better | 0 | 0
  Baseline, Erection ability, Much Better | 1 | 1
  Baseline, Erection ability, A Little Better | 1 | 1
  Baseline, Erection ability, No change | 54 | 55
  Baseline, Erection ability, A Little Worse | 3 | 1
  Baseline, Erection ability, Much worse | 0 | 0
  Baseline, Erection ability, Very Much Worse | 0 | 0
  Baseline, Sexual life, Very Much Better | 0 | 0
  Baseline, sexual life, Much Better | 1 | 1
  Baseline, sexual life, A Little Better | 1 | 0
  Baseline, sexual life, No change | 55 | 56
  Baseline, sexual life, A Little Worse | 2 | 1
  Baseline, sexual life, Much worse | 0 | 0
  Baseline, sexual life, Very Much Worse | 0 | 0
  DB week 24, Erection ability, Very Much Better | 1 | 0
  DB week 24, Erection ability, Much Better | 0 | 0
  DB week 24, Erection ability, A Little Better | 2 | 4
  DB week 24, Erection ability, No change | 49 | 40
  DB week 24, Erection ability, A Little Worse | 5 | 7
  DB week 24, Erection ability, Much worse | 0 | 1
  DB week 24, Erection ability, Very Much Worse | 0 | 0
  DB week 24, Sexual life, Very Much Better | 1 | 0
  DB week 24, sexual life, Much Better | 0 | 1
  DB week 24, sexual life, A Little Better | 3 | 2
  DB week 24, sexual life, No change | 47 | 39
  DB week 24, sexual life, A Little Worse | 6 | 9
  DB week 24, sexual life, Much worse | 0 | 1
  DB week 24, sexual life, Very Much Worse | 0 | 0

58. Secondary Outcome: Change From Baseline in Participants Perception of Sexual Function Measured by Responses to the Global Assessment Questions Open-label Treatment Period
Description: The global assessment questions consist of 2 questions, recording how much the participant perceives his sexual life has changed and how he perceives his ability to achieve and maintain erections has changed, compared to how it was before he began receiving treatment in this study. The wording of these questions were based on the Patient Global Impression of Improvement questionnaire, which was validated for use in the assessment of improvement in stress urinary incontinence. The questions were scored on a 7-point scale.The Baseline assessment was defined as the latest assessment on or before the OL treatment start.
Time Frame: Baseline and up to Week 24
Population: open-label period population
Measure: Number; unit: Participants
Arm/Group | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Number analyzed (Participants) | 49 | 48
Participants
  OL Baseline, Erection ability, Very Much Better | 1 | 0
  OL Baseline, Erection ability, Much Better | 0 | 0
  OL Baseline, Erection ability, A Little Better | 1 | 4
  OL Baseline, Erection ability, No change | 42 | 39
  OL Baseline, Erection ability, A Little Worse | 5 | 5
  OL Baseline, Erection ability, Much worse | 0 | 0
  OL Baseline, Erection ability, Very Much Worse | 0 | 0
  OL Baseline, Sexual life, Very Much Better | 1 | 0
  OL Baseline, sexual life, Much Better | 0 | 1
  OL Baseline, sexual life, A Little Better | 2 | 2
  OL Baseline, sexual life, No change | 40 | 39
  OL Baseline, sexual life, A Little Worse | 6 | 6
  OL Baseline, sexual life, Much worse | 0 | 0
  OL Baseline, sexual life, Very Much Worse | 0 | 0
  OL week 24, Erection ability, Very Much Better | 0 | 0
  OL week 24, Erection ability, Much Better | 2 | 0
  OL week 24, Erection ability, A Little Better | 1 | 4
  OL week 24, Erection ability, No change | 35 | 37
  OL week 24, Erection ability, A Little Worse | 6 | 5
  OL week 24, Erection ability, Much worse | 0 | 0
  OL week 24, Erection ability, Very Much Worse | 0 | 0
  OL week 24, Sexual life, Very Much Better | 0 | 0
  OL week 24, sexual life, Much Better | 2 | 1
  OL week 24, sexual life, A Little Better | 1 | 2
  OL week 24, sexual life, No change | 37 | 39
  OL week 24, sexual life, A Little Worse | 4 | 4
  OL week 24, sexual life, Much worse | 0 | 0
  OL week 24, sexual life, Very Much Worse | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious Adverse Events (AEs) were collected from the start of study medication until follow-up (up to 54 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for Safety Population.
Arm/Group | Placebo (DB) | Dutasteride 0.5 mg (DB) | Placebo (DB)/Dutasteride 0.5 mg (OL) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) | Combined: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL)
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/58 | 1/49 | 0/48 | 1/48
Other Adverse Events (participants affected / at risk) | 5/59 | 10/58 | 1/49 | 4/48 | 13/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (DB) (N=59) | Dutasteride 0.5 mg (DB) (N=58) | Placebo (DB)/Dutasteride 0.5 mg (OL) (N=49) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) (N=48) | Combined: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) (N=48)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (DB) (N=59) | Dutasteride 0.5 mg (DB) (N=58) | Placebo (DB)/Dutasteride 0.5 mg (OL) (N=49) | Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) (N=48) | Combined: Dutasteride 0.5 mg (DB)/Dutasteride 0.5 mg (OL) (N=48)
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 7 | 1 | 0 | 7
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.